CLINICAL TRIAL: NCT05419219
Title: Effectiveness of Multi-domain Tai Chi Digital Therapy for Survivors Affected by the Sequelae of Covid-19 (TaiChi-DTx and Long Covid)
Brief Title: TaiChi-DTx for Treating Long Covid Symptoms
Acronym: TaiChi-DTx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tim Shi (Other)
Responsible Party: Sponsor-Investigator, Tim Shi, Director, GlobalMD Organization Network Corp
Organization: GlobalMD Organization Network Corp (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TaiChi-DTx_for Long Covid
Record Dates: First submitted 2022-05-03; First posted 2022-06-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Fatigue; Dyspnea; Cognitive Impairment; Muscle Pain
Keywords: Long Covid, Tai Chi, Digital Therapeutics
MeSH Terms: conditions — Fatigue; Dyspnea; Cognitive Dysfunction; Myalgia; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: To evaluate the effectiveness of Multi-domain Tai Chi Digital Therapy for treating the long term sequalae symptoms among COVID-19 survivors compared with traditional Tai Chi exercise only as control.
Who Masked: Participant
Masking Description: The Multi-domain Tai Chi-DTx will be provided via a tablet or smart phone. The traditional Tai Chi exercise with background music and respiratory control exercise with 18 BPM metronome, and 40 Hz sound stimulation will be comprised in a 4-week therapeutic session.
  A control arm will be designed in this study, which will use the same way to deliver traditional Tai Chi exercise with plain music background only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- The Multi-domain Tai Chi Digital Therapy Group (Active Comparator): participants will be provided via a tablet or smart phone the traditional Tai Chi exercise with background music and respiratory control exercise with 18 BPM metronome, and 40 Hz sound stimulation for 4-week therapeutic session.
  Interventions: Device: the multi-domain Tai Chi Digital therapy Software Application
- The regular Tai Chi Exercise Group (Placebo Comparator): participants will be provided by the same way to deliver traditional Tai Chi exercise with plain music background, but without respiratory control exercise or 40 Hz sound stimulation. All participants will receive any other routine care or treatment as usual (TAU).
  Interventions: Device: the multi-domain Tai Chi Digital therapy Software Application

INTERVENTIONS:
Device: the multi-domain Tai Chi Digital therapy Software Application — regular Tai Chi exercise, 40 Hz gamma sound stimulation and 18 BPM breath control exercise

SUMMARY:
The randomized controlled trial will be conducted to evaluate the effectiveness of a Multi-domain Tai Chi Digital Therapy for treating the individuals suffering from the long term COVID-19 syndrome (Long COVID).

DETAILED DESCRIPTION:
The randomized controlled trial will be conducted to evaluate the effectiveness of a Multi-domain Tai Chi Digital Therapy for treating the individuals suffering from the long term COVID-19 syndrome (Long COVID).

This intervention will comprise of traditional Tai Chi physical therapy with background music entraining 40 Hz sound wave and respiratory control training. The Multi-domain Tai Chi Digital Therapy will be delivered via a tablet or smart phone to participants for a 4-week therapeutic cycle. Clinical standardized physical tests and self-scored questionnaires will be collected to understand the change in symptoms, including fatigue, dyspnea, and brain fog, as well as absenteeism.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis with SARS-CoV2 infection via PCR during the past 3 to 6 months
2. Must be Grade 2 and Grade 3 assessed by the Post-COVID-19 Functional Status (PCFS) Scale

Exclusion Criteria:

1. Admitted in the Intensive Care Unit due to SARS-COV2 infection or any other serve illness
2. Psychiatric diseases and somatic co-morbidities
3. COVID-19 infections or co-morbidities started or exacerbated during the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity ability measured by 6-minute walking distance measurement (6MWT) | 4 weeks
  The 6-min walk test (6 MWT), a recognized norm by American Thoracic Society, is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-min walk distance (6 MWD) in a 30 meter or 100 foot walkway provides a measure for the integrated response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Overall respiratory relief measured by the Post-COVID-19 Functional Status (PCFS) Scale | 4 weeks
  The PCFS scale covers the entire range of functional limitations, including changes in lifestyle, sports, and social activities, and has been widely used as a standard tool to assess recovery after COVID-19 infections (Garout, M.A, 2022). The assignment of a PCFS scale grade concerns the average situation of the past week. The symptoms included in PCFS are dyspnea, pain, fatigue, muscle weakness, memory loss, depression, and anxiety.
Cognitive impairment improvement measured by the well-validated neuropsychological measurement tests | 4-6 weeks
  Assessment tools including Number Span forward (attention) and backward (working memory) (Becker et al. 2021), and Trail Making Test (processing speed and executive functioning), etc (Douaud, G, et al. 2022).

SECONDARY OUTCOMES:
Change in number of hours/days absent from work related to Long COVID symptoms survey by web-based questionnaires (time frame 6 months after SARS-CoV-2 infection) | 4-6 weeks
  The Symptom Burden Questionnaire™ for Long COVID (SBQ™-LC)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Shi, MD, PhD, Principal Investigator — GlobalMD Organization
Locations (1):
- Tim Shi, Ellicott City, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
the multi-domain Tai Chi Digital Therapy for Long Covid survivors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 12 months
Access Criteria: the public

REFERENCES:
- [Background] Castro JP, Kierkegaard M, Zeitelhofer M. A Call to Use the Multicomponent Exercise Tai Chi to Improve Recovery From COVID-19 and Long COVID. Front Public Health. 2022 Feb 28;10:827645. doi: 10.3389/fpubh.2022.827645. eCollection 2022. PMID 35296042
- [Background] Gaber TAK, Ashish A, Unsworth A. Persistent post-covid symptoms in healthcare workers. Occup Med (Lond). 2021 Jun 16;71(3):144-146. doi: 10.1093/occmed/kqab043. PMID 33830208
- [Background] Groff D, Sun A, Ssentongo AE, Ba DM, Parsons N, Poudel GR, Lekoubou A, Oh JS, Ericson JE, Ssentongo P, Chinchilli VM. Short-term and Long-term Rates of Postacute Sequelae of SARS-CoV-2 Infection: A Systematic Review. JAMA Netw Open. 2021 Oct 1;4(10):e2128568. doi: 10.1001/jamanetworkopen.2021.28568. PMID 34643720
- [Result] Verger A, Kas A, Dudouet P, Goehringer F, Salmon-Ceron D, Guedj E. Visual interpretation of brain hypometabolism related to neurological long COVID: a French multicentric experience. Eur J Nucl Med Mol Imaging. 2022 Jul;49(9):3197-3202. doi: 10.1007/s00259-022-05753-5. Epub 2022 Mar 23. PMID 35320385